CLINICAL TRIAL: NCT04507308
Title: Real-time Experiences With Sleep Training Study
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Erin Kaufman, Assistant Professor of Psychology, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115454
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Borderline Personality Disorder; Sleep Disturbance
Keywords: ecological momentary assessment; electroencephalogram; Transdiagnostic Sleep and Circadian Intervention Youth
MeSH Terms: conditions — Borderline Personality Disorder; Parasomnias

STUDY DESIGN:
Intervention Model Description: All participants are completing the same study procedure.
Masking Description: All participants are completing the same study procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transdiagnostic Sleep and Circadian Intervention (Experimental): All participants will undergo baseline assessment and then complete a brief, single-session sleep-focused intervention based on psychoeduation and handouts from the Youth version of the Transdiagnostic Sleep and Circadian Intervention (TranS-C-Youth).
  Interventions: Behavioral: Single-session sleep intervention drawn from principles of the TranS-C youth protocol

INTERVENTIONS:
Behavioral: Single-session sleep intervention drawn from principles of the TranS-C youth protocol — We are providing participants psychoeducation on sleep and will be going over several handouts from the Youth version of the Transdiagnostic Sleep and Circadian Intervention (TranS-C-Youth) to improve sleep.

SUMMARY:
Borderline personality disorder (BPD) is a serious mental illness that often first emerges in adolescence. Effective treatments are typically expensive, lengthy, and intense (e.g., Dialectical Behavior Therapy). Thus, setting individuals up for treatment success is extremely important. Disrupted sleep is closely linked to many BPD symptoms (e.g., moodiness, impulsivity, interpersonal problems), and people with BPD have a range of sleep-related problems. Importantly, sleep problems may make BPD symptoms worse, longer lasting, and also interfere with learning new skills in treatment. Understanding sleep problems in BPD may help create better interventions, as most therapies for BPD do not currently address sleep difficulties. Although approaches like Cognitive Behaviour Therapy for insomnia (CBT-I) and the Youth version of the Transdiagnostic Sleep and Circadian Intervention (TranS-C-Youth) work well with many populations, scientists don't yet know if youth with BPD features can tolerate a sleep-focused intervention. The investigators will recruit youth between ages 13 and 18 who have 3 or more clinically impairing BPD symptoms from the London community and via clinician referrals. They will also recruit a parent to report on their child's sleep patterns, mental health symptoms, and accompany youth to an intervention session. Participants will complete diagnostic interviews and a range of surveys to assess their current functioning (e.g., sleep, mental health, BPD symptoms). Investigators will also ask youth to report on their BPD symptoms multiple times per day in real time and track their sleep at night for a 10-day period. Participants will also wear a headband to track their brain waves while they sleep. After an initial 10-day monitoring period, youth participants will receive a brief, single-session sleep intervention with their parent using materials from the TranS-C-Youth protocol. Adolescents will be asked to follow a sleep plan created during their visit for three weeks before completing another 10 days of assessment. Participants will complete a follow-up survey battery upon completion of the second real-time survey protocol, and also be invited to complete surveys one-month post intervention. The investigators hypothesize that day-to-day variability in sleep will influence BPD symptom presentation, and vice versa. They also hypothesize that our intervention will improve sleep quantity/quality among an at-risk sample, and may be associated with decreased BPD symptoms relative to baseline.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a persistent and profoundly impairing mental disorder characterized by interpersonal turmoil, severe emotion dysregulation, and impulsivity(1). BPD often first manifests in adolescence(2) and even subthreshold levels of symptoms are associated with significant psychosocial morbidity(3). Approximately 69% to 80% of persons with this condition engage in self-injurious behavior, and as many as 9% die by suicide(4-5). Although efficacious treatment approaches have been developed (e.g., Dialectical Behavior Therapy [DBT];6), they are typically expensive, lengthy, and intensive. Identifying methods for optimizing BPD treatment and prevention is an urgent public health priority.

Disrupted sleep is closely linked to defining characteristics of BPD such as higher sensitivity and reactivity to stress, behavioral impulsivity, interpersonal dysfunction, and poor emotion regulation(7). Studies have documented a range of sleep disturbances among BPD samples, and demonstrated that sleep problems are not better accounted for by concomitant depression or other psychiatric disorders(7-9). Importantly, sleep problems may worsen BPD symptom course and chronicity(10-11), heighten risk of suicide(12-13) and self-harm(14), and interfere with cognitive processes that are vital to behavioral intervention (e.g., memory consolidation, and attentional processes; 15). A greater understanding of sleep disturbance in BPD may help enrich treatment protocols, which currently place limited emphasis on sleep difficulties(11). Although approaches like Cognitive Behaviour Therapy for insomnia (CBT-I) and the Youth version of the Transdiagnostic Sleep and Circadian Intervention (TranS-C-Youth) are effective with many populations(16), it is currently unknown whether sleep-focused interventions can be tolerated or followed adherently by youth with BPD features (who are often extremely dysregulated across affective, interpersonal, and behavioral domains).

Objectives: 1) To assess transactional relations of sleep, interpersonal stressors, affect, impulsive behaviors, and self-harm among youth with BPD features (N = 50); 2) To assess the effects of a brief sleep intervention on subsequent sleep quality (primary outcome) and BPD symptoms (secondary outcome). This pilot study will establish recruitment feasibility, determine the acceptability and efficacy of a sleep-focused intervention among adolescents with BPD features, and provide crucial preliminary data to support future grants.

Methodology. The investigators will use a pre-post intervention design with 2 assessments. Changes in BPD symptoms, self-reported sleep quality, and ambulatory monitoring of electroencephalogram (EEG) during sleep, will be assessed approximately 30 days post-treatment. Two 10-day EMA protocols (one prospective and one post-intervention) will provide data for transactional analyses.

Participants: Adolescents ages 13-18 (N=50) will participate with a parent.

Recruitment will be conducted through physician and therapist referrals and ethics-approved media advertisements and fliers posted in waiting rooms where youth with BPD are likely to be treated (e.g., children's hospital), and common community venues (coffee shops, libraries, community centers). Interested participants (and a parent) will complete a brief telephone screen to determine initial eligibility and schedule two virtual visits.

Research Protocol:

1. Phone Screening/Eligibility:

   * Parental verbal consent for phone screen and Youth verbal assent for phone screen
   * Brief interview to determine eligibility: McLean Screening Interview
   * Schedule virtual visit 1 via Zoom over phone, or during email follow-up
2. Send consent/assent documents via email (forms sent for electronic signature; see "Parental Permission and Authorization Document" and "Assent")

   Consent forms are signed/returned electronically.
3. Baseline Questionnaires:

   - Send parents and youth measures via email for electronic completion:

   Youth questionnaires:
   * Demographic Questionnaire
   * The Difficulties in Emotion Regulation Scale Short Form (DERS-SF)
   * Adolescent Sleep Hygiene Scale
   * Borderline Personality Features Scale for Children-11(BPFS-C-11)
   * PROMIS Pediatric Sleep Disturbances SF8
   * PROMIS Pediatric Sleep Related Impairment SF8
   * Self-Concept and Identity Measure (SCIM)
   * Adolescent Sleep Wake Scale - 10 item version
   * Urgency, Premeditation (lack of), Perseverance (lack of), Sensation Seeking, Positive Urgency, Impulsive Behavior Scale Short form (UPPS-P)
   * Items from the Sleep Practices and Attitudes Questionnaire

   Parent-Report (can be completed online post-visit if needed):
   * Demographic Questionnaire
   * PROMIS Pediatric Sleep Disturbances Parent Proxy SF8
   * PROMIS Pediatric Sleep Practices Parent Proxy
   * Sleep Disturbance Scale for Children
   * PROMIS Pediatric Sleep Related Impairment Parent Proxy SF4
   * Child Behavior Checklist (CBCL)
4. Virtual Visit 1 via Zoom

   * Pre-visit risk assessment with youth
   * Interviews:

     * The Childhood Interview for Borderline Personality Disorder
     * Lifetime Suicide Attempt Self-Injury Interview (L-SASSI)
   * Schedule Sleep Band pick-up over the phone-participants to pick up on campus or coordinate other arrangements, as needed (e.g., mail).
   * Provide psychoeducation and instructions on wearing sleep band and completing EMA protocol
   * End-of-visit risk assessment with youth

     * Participants receive/pick-up sleep band ~
5. Ecological momentary assessment (EMA) and EEG Protocol 1 (10 days):

   * EMA assessments will be collected 5 times per day. Upon waking, participants will report bed time and wake time for calibration with sleep EEG data
   * Each daily survey will assess current mood, sleep, and BPD symptoms since the last prompt (e.g., perceived emotional control/dyscontrol, emotional lability, interpersonal conflict, impulsive behavior, dissociation, self-harm urges/behaviors; see attached EMA protocol).

     * Research staff will monitor EMA responses each morning.
     * When responses during the EMA protocol indicate imminent risk of suicide or self-injury (see EMA protocol for specific rules), the CMHA Ontario's suicide crisis number will automatically display on participants' smart phone, and research staff will immediately receive an automated e-mail. Research staff are able to log into the secure database to view participants' responses, and Dr. Kaufman may contact the participant by telephone for risk assessment and safety planning. Appropriate intervention or follow-up care will be arranged. In cases of immediate safety risk, the research team will define a feasible safety plan with the participant (this may include other members in the participants' network and/or crisis intervention services and emergency care). If child abuse or neglect is disclosed, the alleged abuse will be reported to local child welfare services and provincial/territorial social service ministries. During the consent process, all participants will be informed of limits to confidentiality and our legal obligations to report dangerous situations.

   EMA protocols of similar duration and assessment frequency have been successfully conducted with individuals at risk for self-harm with excellent participant compliance rates (21-23).
6. Call participant to schedule sleep band drop-off (on campus)

   ~ Participant returns sleep band ~
7. Virtual visit 2 via Zoom

   * Pre-visit risk assessment
   * Together, youth and parent watch a video providing psychoeducation about sleep
   * Youth will receive a sleep-focused skills training session with their parent:

     ~A clinical psychology graduate student will complete the following handouts from the TranS-C Youth protocol (an established, evidence-based sleep intervention for adolescents) in collaboration with the participant and their parent:
     * "Case Conceptualization"
     * "Improving Your Sleep Summary"
     * "Rise-up checklist"
     * "Wind-down handout"
     * "Stimulus Control"
     * "My Sleep Goals"
   * Participants will be asked to practice the skills they have learned for the following month and be provided digital copies of their worksheets to support their unique sleep plan.
   * End-of-visit risk assessment

     * 2-week period where youth implement and get accustomed to their new sleep plan ~
8. Call participant to schedule second sleep band pick-up (on campus)

   ~ Participants receive/pick-up sleep band (pick-up within 1 week of call) ~
9. Post-EMA and EEG Protocol 2 (10 days; 3 weeks post-intervention)

   - EMA assessments will proceed as they did for protocol 1 (i.e., 5 times per day), with additional prompts to assess sleep plan/skill usage.
   * Research staff will monitor EMA responses by examining data each morning.
   * When responses during the EMA protocol indicate imminent risk of suicide or self-injury, the CMHA Ontario's suicide crisis number will automatically display on participants' smart phone, and research staff will immediately receive an automated e-mail. Research staff are able to log into the secure database to view participants' responses, and Dr. Kaufman may contact the participant by telephone for risk assessment and safety planning. Appropriate intervention or follow-up care will be arranged. In cases of immediate safety risk, the research team will define a feasible safety plan that includes other members in the participants' network and/or crisis intervention services and emergency care. If child abuse or neglect is disclosed, the alleged abuse will be reported to local child welfare services and provincial/territorial social service ministries. During the consent process, all participants will be informed of limits to confidentiality and our legal obligations to report dangerous situations.
10. Post-test Questionnaires:

    - Send parents and youth measures via email for electronic completion:

    Youth:
    * DERS-SF
    * Adolescent Sleep Hygiene Scale
    * BPFS-C-11
    * PROMIS Pediatric Sleep Disturbances SF8
    * PROMIS Pediatric Sleep Related Impairment SF8
    * SCIM
    * Adolescent Sleep Wake Scale - 10 item version
    * UPPS-P
    * Items from the Sleep Practices and Attitudes Questionnaire

    Parents:
    * PROMIS Pediatric Sleep Disturbances Parent Proxy SF8
    * PROMIS Pediatric Sleep Practices Parent Proxy
    * Sleep Disturbance Scale for Children
    * PROMIS Pediatric Sleep Related Impairment Parent Proxy SF4 ~Questionnaires need to be completed no later than 1 week after 2nd EMA protocol.~
11. Call participant to schedule sleep band drop-off (on campus) Participant drops-off sleep band
12. Payment given for EMA electronically (emailed) after sleep band is returned undamaged
13. 1-Month Follow-up

    * Participants will be emailed questionnaires 1-month following completion of their second EMA protocol. Those who complete these questionnaires will be entered to win a drawing for a $50 gift card (one for parents and one for teens)
    * Youth emailed:

      * DERS-SF
      * Adolescent Sleep Hygiene Scale
      * BPFS-C-11
      * PROMIS Pediatric Sleep Disturbances SF8
      * PROMIS Pediatric Sleep Related Impairment SF8
      * SCIM
      * Adolescent Sleep Wake Scale - 10 item version
    * Parents emailed:

      * PROMIS Pediatric Sleep Disturbances Parent Proxy SF8
      * PROMIS Pediatric Sleep Practices Parent Proxy
      * Sleep Disturbance Scale for Children
      * PROMIS Pediatric Sleep Related Impairment Parent Proxy SF4

ELIGIBILITY:
Inclusion Criteria:

* Youth between 13 and 18 years of age
* 3+ clinically impairing symptoms of borderline personality disorder as determined via screening interview
* Parent available to complete informant-report and accompany participant to sleep intervention session
* Participant has a cellular phone or reliable access to a computer to complete ecological momentary assessment protocol

Exclusion Criteria:

* Participants without English language proficiency will be excluded as the study requires verbal and written components delivered exclusively in English.
* Participants with fewer than 3 clinically impairing BPD symptoms will be excluded from the study.
* We will exclude adolescents who present with an intellectual disability or have a schizophrenia spectrum diagnosis.
* Participants who do not have a parent/caregiver available to attend the virtual intervention session will also be excluded from the study.
* Participants without access to a personal cellular phone or reliable access to a computer with internet will be excluded.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Sleep improvement | Baseline data will be collected over the course of a 10 day period (including ecological momentary assessment data) and compared to data collected over a second 10 day window one-month post intervention.
  Change from baseline sleep data (self- and informant-report, electroencephalogram data during sleep, and ecological momentary assessment data) to post-intervention data.
Change in borderline personality disorder symptoms | Baseline data will be collected over the course of a 10 day period (including ecological momentary assessment data) and compared to data collected over a second 10 day window one-month post intervention.
  Change in participants' BPD symptoms from baseline (assessed via diagnostic interview and a 10-day ecological momentary assessment protocol) to one-month post-intervention (via a second 10-day ecological momentary assessment protocol).

CONTACTS AND LOCATIONS:
Overall Officials: Erin A Kaufman, Ph.D., Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario Westminster Hall, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with scientific collaborators in the future. Given the sensitive nature of study data, and that our sample includes vulnerable youth recruited from the London area, we will not provide unrestricted access to all study variables. A subset of de-identified questionnaire, interview, and psychophysiological data may be made available by request. Researchers interested in more sensitive data (e.g., demographic variables that, in combination, could increase the odds of participant identification [age, sex, race, ethnicity, gender identity, and sexual orientation]) can request variables of interest from the principle investigator, and will be asked to complete a plan for data security.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Each of the above supporting information may be provided following the end of the study and publication of primary findings. Directly or indirectly identifiable data will be destroyed after 7 years (consistent with University of Western Ontario's policy). All other data will be available for 25 years.
Access Criteria: Interested researchers can email the principle investigator to request de-identified data. They will be asked to provide a plan for data security.

REFERENCES:
- [Background] American Psychiatric Association, & American Psychiatric Association. DSM-5 Task Force. (2013). Diagnostic and statistical manual of mental disorders: DSM-5. (Fifth edition.). Washington, DC: American Psychiatric Association.
- [Background] Kaess M, Brunner R, Chanen A. Borderline personality disorder in adolescence. Pediatrics. 2014 Oct;134(4):782-93. doi: 10.1542/peds.2013-3677. Epub 2014 Sep 22. PMID 25246626
- [Background] Zimmerman M, Chelminski I, Young D, Dalrymple K, Martinez J. Is dimensional scoring of borderline personality disorder important only for subthreshold levels of severity? J Pers Disord. 2013 Apr;27(2):244-51. doi: 10.1521/pedi.2013.27.2.244. PMID 23514187
- [Background] Soloff PH, Lis JA, Kelly T, Cornelius J, Ulrich R. Risk factors for suicidal behavior in borderline personality disorder. Am J Psychiatry. 1994 Sep;151(9):1316-23. doi: 10.1176/ajp.151.9.1316. PMID 8067487
- [Background] Zanarini MC, Frankenburg FR, Hennen J, Reich DB, Silk KR. The McLean Study of Adult Development (MSAD): overview and implications of the first six years of prospective follow-up. J Pers Disord. 2005 Oct;19(5):505-23. doi: 10.1521/pedi.2005.19.5.505. PMID 16274279
- [Background] Linehan, M. M. (1993). Cognitive-behavioral treatment of borderline personality disorder. New York: Guilford Press.
- [Background] Winsper C, Tang NK, Marwaha S, Lereya ST, Gibbs M, Thompson A, Singh SP. The sleep phenotype of Borderline Personality Disorder: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2017 Feb;73:48-67. doi: 10.1016/j.neubiorev.2016.12.008. Epub 2016 Dec 15. PMID 27988314
- [Background] Bastien CH, Guimond S, St-Jean G, Lemelin S. Signs of insomnia in borderline personality disorder individuals. J Clin Sleep Med. 2008 Oct 15;4(5):462-70. PMID 18853705
- [Background] Benson KL, King R, Gordon D, Silva JA, Zarcone VP Jr. Sleep patterns in borderline personality disorder. J Affect Disord. 1990 Apr;18(4):267-73. doi: 10.1016/0165-0327(90)90078-m. PMID 2140379
- [Background] Plante DT, Frankenburg FR, Fitzmaurice GM, Zanarini MC. Relationship between sleep disturbance and recovery in patients with borderline personality disorder. J Psychosom Res. 2013 Apr;74(4):278-82. doi: 10.1016/j.jpsychores.2013.01.006. Epub 2013 Feb 11. PMID 23497827
- [Background] Selby, E.A., Ribeiro, J.D., Joiner Jr., T.E. (2013). What dreams may come: Emotional cascades and nightmares in borderline personality disorder. Dreaming, 23, 126.
- [Background] Balestrieri M, Rucci P, Sbrana A, Ravani L, Benvenuti A, Gonnelli C, Dell'osso L, Cassano GB. Lifetime rhythmicity and mania as correlates of suicidal ideation and attempts in mood disorders. Compr Psychiatry. 2006 Sep-Oct;47(5):334-41. doi: 10.1016/j.comppsych.2006.01.004. Epub 2006 Apr 21. PMID 16905394
- [Background] Winsper C, Tang NK. Linkages between insomnia and suicidality: prospective associations, high-risk subgroups and possible psychological mechanisms. Int Rev Psychiatry. 2014 Apr;26(2):189-204. doi: 10.3109/09540261.2014.881330. PMID 24892894
- [Background] Semiz UB, Basoglu C, Ebrinc S, Cetin M. Nightmare disorder, dream anxiety, and subjective sleep quality in patients with borderline personality disorder. Psychiatry Clin Neurosci. 2008 Feb;62(1):48-55. doi: 10.1111/j.1440-1819.2007.01789.x. PMID 18289141
- [Background] Curcio G, Ferrara M, De Gennaro L. Sleep loss, learning capacity and academic performance. Sleep Med Rev. 2006 Oct;10(5):323-37. doi: 10.1016/j.smrv.2005.11.001. Epub 2006 Mar 24. PMID 16564189
- [Background] Essner B, Noel M, Myrvik M, Palermo T. Examination of the Factor Structure of the Adolescent Sleep-Wake Scale (ASWS). Behav Sleep Med. 2015;13(4):296-307. doi: 10.1080/15402002.2014.896253. Epub 2014 Apr 17. PMID 24742264
- [Background] LeBourgeois MK, Giannotti F, Cortesi F, Wolfson AR, Harsh J. The relationship between reported sleep quality and sleep hygiene in Italian and American adolescents. Pediatrics. 2005 Jan;115(1 Suppl):257-65. doi: 10.1542/peds.2004-0815H. PMID 15866860
- [Background] Harvey, A.G., 2015. A transdiagnostic intervention for youth sleep and circadian problems. Cognitive and Behavioral Practice, 3, 341-355.
- [Background] Bastida-Pozuelo MF, Sanchez-Ortuno MM, Meltzer LJ. Nurse-led brief sleep education intervention aimed at parents of school-aged children with neurodevelopmental and mental health disorders: Results from a pilot study. J Spec Pediatr Nurs. 2018 Oct;23(4):e12228. doi: 10.1111/jspn.12228. Epub 2018 Nov 27. PMID 30480370
- [Background] Ellis JG, Cushing T, Germain A. Treating Acute Insomnia: A Randomized Controlled Trial of a "Single-Shot" of Cognitive Behavioral Therapy for Insomnia. Sleep. 2015 Jun 1;38(6):971-8. doi: 10.5665/sleep.4752. PMID 25515106
- [Background] Husky M, Olie E, Guillaume S, Genty C, Swendsen J, Courtet P. Feasibility and validity of ecological momentary assessment in the investigation of suicide risk. Psychiatry Res. 2014 Dec 15;220(1-2):564-70. doi: 10.1016/j.psychres.2014.08.019. Epub 2014 Aug 15. PMID 25155939
- [Background] Jahng S, Wood PK, Trull TJ. Analysis of affective instability in ecological momentary assessment: Indices using successive difference and group comparison via multilevel modeling. Psychol Methods. 2008 Dec;13(4):354-75. doi: 10.1037/a0014173. PMID 19071999
- [Background] Trull TJ, Solhan MB, Tragesser SL, Jahng S, Wood PK, Piasecki TM, Watson D. Affective instability: measuring a core feature of borderline personality disorder with ecological momentary assessment. J Abnorm Psychol. 2008 Aug;117(3):647-61. doi: 10.1037/a0012532. PMID 18729616